CLINICAL TRIAL: NCT01220518
Title: Randomized, Double-blind, Parallel-group, Phase 1 Study
Brief Title: Program evaLuating the Autoimmune Disease iNvEstigational Drug cT-p13 in AS Patients(PLANETAS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT-P13 1.1
Record Dates: First submitted 2010-10-04; First posted 2010-10-14 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT-P13 (Active Comparator): infliximab
  Interventions: Drug: Infliximab
- Remicade (Active Comparator): infliximab
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Infliximab 5mg/kg is going to be administered for both arm as a 2-hour infusion per dose.

SUMMARY:
This study is the trial to demonstrate how our product is similar to remicade by comparing the results of blood samples in active Ankylosing Spondylitis patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with active ankylosing spondylitis
* BASDAI score ≥ 4 and visual analogue scale(VAS) score of spinal pain ≥ 4

Exclusion Criteria:

* have total ankylosing of spine
* have allergies to infliximab
* serious infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
PK equivalence to remicade | PK sampling at week 22

SECONDARY OUTCOMES:
Proportion of patients achieving clinical response according to the Assessment of SpondyloArthritis International Society (ASAS) 20% criteria | at week 14, 30 and 54
Proportion of patients achieving clinical response according to the Assessment of SpondyloArthritis International Society (ASAS) 40 criteria | at week 14, 30 and 54
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Weeks 14, 30 and 54 compared with Baseline | at week 14, 30 and 54
Bath Ankylosing Spondylitis Functional Index (BASFI) at Weeks 14, 30 and 54 compared with Baseline | at week 14, 30 and 54
Bath Ankylosing Spondylitis Metrology Index (BASMI) at Weeks 14, 30 and 54 compared with Baseline | at weeks 14, 30 and 54
Chest expansion at Weeks 14, 30 and 54 compared with Baseline | at weeks 14, 30 and 54
Quality of life questionnaire (SF-36) | at week 14, 30 and 54

CONTACTS AND LOCATIONS:
Overall Officials: Won Park, M.D., Ph.D., Principal Investigator — Inha University Hospital
Locations (1):
- Inha University Hostpital, Incheon, South Korea

REFERENCES:
- [Derived] Eser A, Reinisch W, Schreiber S, Ahmad T, Boulos S, Mould DR. Increased Induction Infliximab Clearance Predicts Early Antidrug Antibody Detection. J Clin Pharmacol. 2021 Feb;61(2):224-233. doi: 10.1002/jcph.1732. Epub 2020 Sep 9. PMID 32905628
- [Derived] Park W, Yoo DH, Jaworski J, Brzezicki J, Gnylorybov A, Kadinov V, Sariego IG, Abud-Mendoza C, Escalante WJ, Kang SW, Andersone D, Blanco F, Hong SS, Lee SH, Braun J. Comparable long-term efficacy, as assessed by patient-reported outcomes, safety and pharmacokinetics, of CT-P13 and reference infliximab in patients with ankylosing spondylitis: 54-week results from the randomized, parallel-group PLANETAS study. Arthritis Res Ther. 2016 Jan 20;18:25. doi: 10.1186/s13075-016-0930-4. PMID 26795209